CLINICAL TRIAL: NCT03668613
Title: A Randomized, Open-label, Multicenter Trial to Assess the Efficacy of Subcutaneous Secukinumab after12 Weeks of Treatment, and to Assess the Long-term Safety, Tolerability, Efficacy in Subjects From 6 to <18 Years of Age With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: Study to Assess the Long-term Safety, Tolerability, Efficacy of Secukinumab in Pediatric Patients of Age 6 to <18 Years, With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAIN457A2311; 2017-004515-39 (EudraCT Number)
Record Dates: First submitted 2018-08-23; First posted 2018-09-12 (Actual); Results first posted 2021-07-23 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Moderate to Severe Chronic Plaque-type Psoriasis
Keywords: pediatric; secukinumab; plaque psoriasis; AIN457A; Skin condition; skin disease; itching condition; psoriasis vulgaris; relapsing/remitting psoriasis; immune-mediated systemic disease; skin lesions; red skin lesions; scaly patches; papules; plaques; itching
MeSH Terms: conditions — Skin Diseases; Recurrence; Plaque, Amyloid; Pruritus | interventions — secukinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- secukinumab low dose (Experimental): secukinumab low dose
  Interventions: Drug: secukinumab low dose
- secukinumab high dose (Experimental): secukinumab high dose
  Interventions: Drug: secukinumab high dose

INTERVENTIONS:
Drug: secukinumab low dose — dose depends on the weight group
  Other Names: AIN457
  Arms: secukinumab low dose
Drug: secukinumab high dose — dose depends on the weight group
  Other Names: AIN457
  Arms: secukinumab high dose

SUMMARY:
This was an open-label, parallel-group, two-arm, multicenter study in pediatric subjects aged 6 years to less than 18 years, at randomization, with moderate to severe chronic plaque psoriasis. 84 subjects (most with moderate severity) were enrolled. Subjects were stratified by weight and disease severity.

DETAILED DESCRIPTION:
This was an open-label, parallel group, two-arm, multi-center, trial in pediatric subjects aged 6 years to less than 18 years, at randomization, with moderate to severe chronic, plaque psoriasis. The study consists of 3 periods: screening (up to 4 weeks), treatment (Week 208) and post-treatment follow-up (Week 224).

Approximately 80 subjects (at least 60 subjects with moderate psoriasis) were planned to be enrolled in about 40 centers worldwide and targeted to have at least 5 subjects in the < 25kg body weight, and at least 10 subjects in each of the other two weight groups (25-< 50 kg and ≥ 50 kg). Adolescents (12-< 18 years) and children (6-< 12 years) were included from the beginning of this study, since the DMC had approved already the enrollment of children (6-< 12 years) in the study CAIN457A2310 (NCT02471144). Subjects received the appropriate dose based on their body weight category.

For the statistical analysis for outcome measures 1 and 2, there was no 'within study' control arm. A historical placebo control was obtained using data from qualifying trials and used as the comparator for the primary and key secondary endpoint analysis. This was in line with the guidance from and discussions with Health Authorities including FDA and EMA (PDCO), which suggested reducing placebo exposure as well as overall clinical trial burden for the pediatric population and accepted an extrapolation approach (EMA 2012). Historical placebo data included in this study were based on clinical appropriateness and alignment of definitions (endpoints, clinical disease population and time point of assessment). Integrated in the analysis were placebo data from Novartis-reported secukinumab adult placebo-controlled studies (CAIN457A2302 (NCT01544595 and NCT01365455), CAIN457A2303 (NCT01544595 and NCT01358578), CAIN457A2308 (NCT01555125) and CAIN457A2309 (NCT01636687)) and pediatric placebo-controlled study CAIN457A2310. In addition, pediatric placebo-controlled study data from the literature on other biologics (e.g. etanercept, ustekinumab) were utilized (Paller et al 2008, Landells et al 2015).

If the subject moved into a higher or lower weight group at two consecutive visits with weight measurements during the maintenance (from Week 12 onwards as assessed at 4 weekly visits or during extension treatment period (as assessed at scheduled site visits), then the subject was dosed according to the new (higher or lower) weight group respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed assent and parental permission (age as per local law) obtained at screening before any assessment is performed.
2. Must be 6 to less than 18 years of age at the time of randomization
3. Moderate to Severe plaque psoriasis, defined as a PASI score ≥ 12, and IGA mod 2011 score of ≥ 3, and BSA involvement of ≥10%, at randomization.
4. Subject being regarded by the investigator to be a candidate for systemic therapy.

Exclusion Criteria:

1. Forms of psoriasis other than chronic plaque-type active at randomization
2. Drug-induced psoriasis
3. Ongoing use of prohibited treatments
4. Female subjects of childbearing potential defined as all women physiologically capable of becoming pregnant, unless they are using effective methods of contraception during dosing and for 16 weeks after stopping study treatment
5. Pregnant or nursing (lactating) females
6. Subjects with total WBC count <2,500/μL, or platelets <100,000/μL or neutrophils <1,500/μL or hemoglobin <8.5 g/dL at screening
7. Previous exposure to secukinumab or any other biologic drug directly targeting IL-17 or the IL-17 receptor

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2019-09-19 (Actual); Study Completion 2023-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (23):
- United States (4):
  - First OC Dermatology, Fountain Valley, California
  - Private Practice, Jacksonville, Florida
  - Novartis Investigative Site, Lebanon, New Hampshire
  - Texas Derm and Laser Specialists ., San Antonio, Texas
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Liège
- Czechia (2):
  - Novartis Investigative Site, Hradec Králové, CZE
  - Novartis Investigative Site, Prague, Prague 1
- Novartis Investigative Site, Tartu, Estonia
- Germany (2):
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Münster
- Novartis Investigative Site, Lima, Peru
- Poland (3):
  - Novartis Investigative Site, Warsaw, Mazowian
  - Novartis Investigative Site, Rzeszów
  - Novartis Investigative Site, Wroclaw
- Russia (4):
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Krasnodar
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
- Spain (4):
  - Novartis Investigative Site, Esplugues de Llobregat, Barcelona
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.
URL: https://clinicalstudydatarequest.com/

REFERENCES:
- [Derived] Kingo K, Papanastasiou P, Beissert S, Lazareva S, Villa AV, Bartonova J, Ballona R, Bansal A, Martin R, Fan H, O'Doherty C, Ravichandran S, Magnolo N. Long-Term Efficacy and Safety of Secukinumab in Children and Adolescents with Moderate-to-Severe Chronic Plaque Psoriasis: Four-Year Results of a Randomized, Phase III, Open-Label Trial. Paediatr Drugs. 2025 Nov;27(6):749-759. doi: 10.1007/s40272-025-00715-4. Epub 2025 Aug 28. PMID 40874954
- [Derived] Sticherling M, Nikkels AF, Hamza AM, Kwong P, Szepietowski JC, El Sayed M, Ghislain PD, Khotko AA, Patekar M, Ortmann CE, Forrer P, Papanastasiou P, Keefe D. Secukinumab in Pediatric Patients with Plaque Psoriasis: Pooled Safety Analysis from Two Phase 3 Randomized Clinical Trials. Am J Clin Dermatol. 2023 Sep;24(5):821-835. doi: 10.1007/s40257-023-00782-8. Epub 2023 Jun 21. PMID 37341961
- [Derived] Magnolo N, Kingo K, Laquer V, Browning J, Reich A, Szepietowski JC, Keefe D, Papanastasiou P, Bao W, Forrer P, Patekar M. Efficacy of Secukinumab Across Subgroups and Overall Safety in Pediatric Patients with Moderate to Severe Plaque Psoriasis: Week 52 Results from a Phase III Randomized Study. Paediatr Drugs. 2022 Jul;24(4):377-387. doi: 10.1007/s40272-022-00507-0. Epub 2022 Jun 13. PMID 35698000
- [Derived] Magnolo N, Kingo K, Laquer V, Browning J, Reich A, Szepietowski JC, Keefe D, Mazur R, Ghelani P, Forrer P, Wraith L, Patekar M. A phase 3 open-label, randomized multicenter study to evaluate efficacy and safety of secukinumab in pediatric patients with moderate to severe plaque psoriasis: 24-week results. J Am Acad Dermatol. 2022 Jan;86(1):122-130. doi: 10.1016/j.jaad.2021.08.066. Epub 2021 Sep 30. PMID 34555481
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2306

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 92 subjects were screened of which 84 subjects completed the screening phase and were randomized to the Secukinumab Low dose and High dose groups in a 1:1 ratio.
Pre-assignment Details: A total of 92 subjects were screened of which 84 subjects completed the screening phase and were randomized to the Secukinumab Low dose and High dose groups in a 1:1 ratio.
Groups:
- AIN457 Low Dose: Subcutaneous (s.c.) secukinumab injections at randomization and weekly until Week 4, thereafter every 4 weeks until Wk 204. Patients received secukinumab 75 mg (if weighing < 50kg) or 150 mg (if weighing >= 50kg)
- AIN457 High Dose: Subcutaneous (s.c.) secukinumab injections at randomization and weekly until Week 4, thereafter every 4 weeks until Wk 204. Patients received secukinumab 75 mg (if weighing < 25kg) or 150mg (if weighing 25 to < 50kg) or 300 mg (if weighing >=50 kg)
Period: Overall Study
Arm/Group | AIN457 Low Dose | AIN457 High Dose
Started | 42 | 42
Completed | 31 | 36
Not Completed | 11 | 6
Not completed — Adverse Event | 1 | 2
Not completed — Lack of Efficacy | 5 | 1
Not completed — Pregnancy | 0 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Guardian decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AIN457 Low Dose | AIN457 High Dose | Total
Number analyzed (Participants) | 42 | 42 | 84
Age, Customized [Number; unit: Participants]
  6 to <12 years | 17 | 16 | 33
  12 to <18 years | 25 | 26 | 51
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 25 | 45
  Male | 22 | 17 | 39
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 39 | 38 | 77
  Black or African American | 1 | 0 | 1
  Asian | 1 | 0 | 1
  American Indian or Alaska Native | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Participants With PASI 75 Response
Description: Psoriasis Area and Severity Index (PASI):Combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72(maximal disease). Body is divided into 4 areas for scoring (head, trunk, upper limbs and lower limbs); each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, Erythema,Thickening (plaque elevation, induration) & Scaling(desquamation). Scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section(head: 0.1, upper limbs: 0.2 body: 0.3 lower limbs: 0.4). Psoriasis Area and Severity Index (PASI) will be assessed/calculated as per standard procedure. PASI 75 represents the percentage (or number)of patients who have achieved a 75% or more reduction in their PASI score from baseline. PASI 100 indicates patients who have achieved a complete resolution of all disease.
Time Frame: Week 12
Population: Full Analysis Set: The FAS comprised all patients from the randomized set to whom study treatment had been assigned
Measure: Count of Participants; unit: Participants
Arm/Group | AIN457 Low Dose | AIN457 High Dose
Number analyzed (Participants) | 42 | 42
Participants | 39 | 39
Statistical Analysis 1: Comparison: AIN457 Low Dose; Compared to historical placebo; Test type: Superiority; Bayesian method using (MAP); Predicted Log-OR = 4.862, 95% CI 2-sided [3.422 to 6.782]
Statistical Analysis 2: Comparison: AIN457 High Dose; Compared to historical placebo; Test type: Superiority; Bayesian method using (MAP); Predicted log-OR = 4.836, 95% CI 2-sided [3.422 to 6.772]

2. Primary Outcome: Number and Percentage of Participants With IGA Mod 2011 0 or 1 Response
Description: Investigator will assess the disease using the validated Investigator Global Assessment (IGA) mod 2011 and rate the disease from a score of 0 (clear skin) to 4 (severe disease)
Time Frame: Week 12
Population: Full Analysis Set: The FAS comprised all patients from the randomized set to whom study treatment had been assigned
Measure: Count of Participants; unit: Participants
Arm/Group | AIN457 Low Dose | AIN457 High Dose
Number analyzed (Participants) | 42 | 42
Participants | 33 | 35
Statistical Analysis 1: Comparison: AIN457 Low Dose; Compared to historical placebo; Test type: Superiority; Bayesian method using (MAP); Predicted log -OR = 4.292, 95% CI 2-sided [2.638 to 6.513]
Statistical Analysis 2: Comparison: AIN457 High Dose; Compared to historical placebo; Test type: Superiority; Bayesian method using (MAP); Predicted log-OR = 4.606, 95% CI 2-sided [2.919 to 6.780]

3. Secondary Outcome: Number and Percentage of Participants With PASI 90 Response
Description: Psoriasis Area and Severity Index (PASI) was assessed/calculated as per the standard procedure.
  PASI 90 represents the percentage (or number) of patients who have achieved a 90% or more reduction in their PASI score from baseline. PASI 100 indicates patients who have achieved a complete resolution of all disease.
Time Frame: Week 12
Population: Full Analysis Set: The FAS comprised all patients from the randomized set to whom study treatment had been assigned
Measure: Count of Participants; unit: Participants
Arm/Group | AIN457 Low Dose | AIN457 High Dose
Number analyzed (Participants) | 42 | 42
Participants | 29 | 32
Statistical Analysis 1: Comparison: AIN457 Low Dose; Test type: Superiority; Bayesian method using (MAP); Predicted log-OR = 4.367, 95% CI 2-sided [2.916 to 6.202]
Statistical Analysis 2: Comparison: AIN457 High Dose; Test type: Superiority; Bayesian method using (MAP); Predicted log-OR = 4.709, 95% CI 2-sided [3.201 to 6.580]

4. Secondary Outcome: Secukinumab Concentration in Serum
Description: Mean (Standard Deviation) Secukinumab concentration levels in serum over time.
Time Frame: Baleine, Weeks 4, 12, 13, 14, 15, 16, 24, 52, 104, 156, 208
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | AIN457 Low Dose | AIN457 High Dose
Number analyzed (Participants) | 42 | 42
mcg/mL
  Baseline | 0.00 (0.00) | 0.00 (0.00)
  Week 4 (n=40,40): number analyzed (Participants) | 40 | 40
  Week 4 (n=40,40) | 74.2 (33.0) | 135 (45.3)
  Week 12 (n=40, 39): number analyzed (Participants) | 40 | 39
  Week 12 (n=40, 39) | 34.8 (10.9) | 69.6 (29.2)
  Week 13 (n=38,33): number analyzed (Participants) | 38 | 33
  Week 13 (n=38,33) | 47.1 (17.4) | 91.2 (34.1)
  Week 14 (n=40, 39): number analyzed (Participants) | 40 | 39
  Week 14 (n=40, 39) | 40.9 (15.5) | 78.4 (29.8)
  Week 15 (n=38,35): number analyzed (Participants) | 38 | 35
  Week 15 (n=38,35) | 34.6 (12.4) | 65.7 (28.9)
  Week 16 (n=40,37): number analyzed (Participants) | 40 | 37
  Week 16 (n=40,37) | 30.9 (11.2) | 55.2 (24.9)
  Week 24 (n=42, 38): number analyzed (Participants) | 42 | 38
  Week 24 (n=42, 38) | 26.0 (10.8) | 48.0 (21.4)
  Week 52 (n=37,38): number analyzed (Participants) | 37 | 38
  Week 52 (n=37,38) | 25.0 (9.01) | 42.7 (17.0)
  Week 104 (n=39,33): number analyzed (Participants) | 39 | 33
  Week 104 (n=39,33) | 21.9 (10.8) | 39.3 (12.1)
  Week 156 (n=34,32): number analyzed (Participants) | 34 | 32
  Week 156 (n=34,32) | 19.3 (8.68) | 35.0 (14.1)
  Week 208 (n=25,28): number analyzed (Participants) | 25 | 28
  Week 208 (n=25,28) | 16.7 (6.25) | 38.8 (17.2)

5. Secondary Outcome: Summary Table of Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a clinical investigation participant after providing written informed consent for participation in the study.
  Treatment emergent adverse events in this study are events that started after the first dose of study treatment and until 84 days after the last study treatment, or events present prior to the first dose of treatment which increased in severity based on preferred term within 84 days after the last study treatment.
Time Frame: Adverse events are reported from the first dose of study-drug until the end of the treatment period (at Week 208) plus 16 weeks additional follow up reporting, for a maximum timeframe of approximately 224 weeks.
Population: Safety set
Measure: Count of Participants; unit: Participants
Arm/Group | AIN457 Low Dose | AIN457 High Dose
Number analyzed (Participants) | 42 | 42
Participants
  Subjects with any AE(s) | 33 | 35
  Subjects with serious or other significant events - Death | 0 | 0
  Subjects with serious or other significant events - Non-fatal SAE(s) | 4 | 2
  Subjects with serious or other significant events - Discontinued study treatment due to any AE(s) | 1 | 2

ADVERSE EVENTS:
Time Frame: Adverse events are reported from the first dose of study-drug until the end of the treatment period (at Week 208) plus 16 weeks additional follow up reporting, for a maximum timeframe of approximately 224 weeks.
Description: Treatment emergent adverse events in this study are events that started after the first dose of study treatment and until 84 days after the last study treatment, or events present prior to the first dose of treatment which increased in severity based on preferred term within 84 days after the last study treatment.
Arm/Group | AIN457 Low Dose | AIN457 High Dose
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/42
Serious Adverse Events (participants affected / at risk) | 4/42 | 2/42
Other Adverse Events (participants affected / at risk) | 30/42 | 27/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 Low Dose (N=42) | AIN457 High Dose (N=42)
Crohn's disease (Gastrointestinal disorders) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 1 | 0
Infectious mononucleosis (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Intentional self-injury (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 Low Dose (N=42) | AIN457 High Dose (N=42)
Leukopenia (Blood and lymphatic system disorders) | 3 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 3
Vomiting (Gastrointestinal disorders) | 3 | 2
Pyrexia (General disorders) | 6 | 1
COVID-19 (Infections and infestations) | 11 | 9
Influenza (Infections and infestations) | 3 | 1
Nasopharyngitis (Infections and infestations) | 13 | 7
Rhinitis (Infections and infestations) | 1 | 3
Tonsillitis (Infections and infestations) | 2 | 4
Upper respiratory tract infection (Infections and infestations) | 0 | 6
Viral upper respiratory tract infection (Infections and infestations) | 1 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Headache (Nervous system disorders) | 3 | 2
Acne (Skin and subcutaneous tissue disorders) | 7 | 2
Eczema (Skin and subcutaneous tissue disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-09-25): https://cdn.clinicaltrials.gov/large-docs/13/NCT03668613/Prot_002.pdf
  • Statistical Analysis Plan (2023-09-27): https://cdn.clinicaltrials.gov/large-docs/13/NCT03668613/SAP_003.pdf